CLINICAL TRIAL: NCT03862209
Title: Large-scale Implementation of Community-based Mental Health Care for People With Severe and Enduring Mental Ill Health in Europe
Brief Title: Community-based Mental Health Care for People With Severe and Enduring Mental Ill Health (RECOVER-E) Croatia
Acronym: RECOVER-E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinički Bolnički Centar Zagreb (Other)
Collaborators: Stichting Trimbos-Instituut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KBC Zagreb RECOVER-E
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Severe Mental Disorder; Schizophrenia; Bipolar Disorder; Severe Depression
Keywords: Community implementation; Community engagement; patient centerednessP; Implementation science; Co-creation; Iterative learning processes
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Two study groups both consisting of patients with SMI (severe mental illness). One group will be receiving care as usual, which in the actual setting means mostly medical treatment, without home care and assertive treatment through community based outreach teams. Another, intervention group, will be receiving assertive treatment care, with mobile assertive teams, consisting of at least three team members.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community mental health team (CMHT) (Experimental): CMHTs will be multidisciplinary; that is, staff will be appointed to the CMHTs that include nurses, social workers, psychiatrists, psychologists, and in this project, a peer expert (a person with lived experience of mental health services). All staff within the CMHT will have defined roles and responsibilities that align with the staff functions, roles and linkages detailed in evidence-based service delivery models for community mental health teams. Participant will randomly be assigned to CMHT that will provide outreach mental health care during the project.
  Interventions: Other: Community mental health team
- Standard care (No Intervention): Health care settings and their providers randomised to the control condition receive usual care: participant will gain standard care; ambulatory care, day hospitals or hospital admission.

INTERVENTIONS:
Other: Community mental health team — CMHT will provide home-based treatment inclusive of crisis resolution services and procedures for early recognition of subclinical psychosis and bipolar disorder, and intensive case management. Integrated care (i.e. health and social care interventions) will be provided to all clients. Furthermore, health and social care evidence-based interventions for severe mental illness (SMI) will be employed during home treatment, such as family-based interventions, motivational interviewing, and cognitive behavioural therapies, combined with medication management and identifying employment (paid and non paid options) and support in finding and maintaining this employment, recovery groups and housing opportunities.
  Other Names: CMHT
  Arms: Community mental health team (CMHT)

SUMMARY:
To contribute to improving the level of functioning and quality of life and mental health outcomes for people with severe and enduring mental ill health (SMI) (schizophrenia, bipolar disorder, depression) by adapting and up scaling the implementation of a community-based service delivery model in Croatia.

DETAILED DESCRIPTION:
For nearly 900 million people living in Europe, mental disorders constitute the most significant yet most neglected public health problem: depression affects an estimated 30.3 million Europeans, and psychotic disorders 5 million Europeans. People with severe and enduring mental ill health want the same things out of life as other citizens but are often placed in a vulnerable position and are hence afforded less opportunities to attain their goals and thus experience a lower quality of life, and have a lower life expectancy compared to the general population. For many countries that have undergone mental health services reform or have health systems in transition, efforts to make such comprehensive community-based mental health services available resulted in short-lived outcomes or are still to demonstrate substantial impact. RECOVER-E's aims to ensure well-functioning community mental health teams in 5 countries in Europe (Macedonia, Romania, Bulgaria, Croatia, and Montenegro), which will serve as the central node for coordination and provision of care for people with SMI. Our project narrows the implementation gap by going beyond infrastructure changes and pursuing the development of human resource capacity and care pathways that can be distilled in a comprehensive pathway to scale for regional and national decision-makers for uptake after the project's life span. RECOVER-E will: 1) Develop evidence based care pathways and treatment protocols for transition to scale for regional and national decision makers in 5 implementation sites; 2) Establish a peer to peer capacity building partnership in community mental health by linking a European expert panel with key stakeholders in 5 implementation sites to co-create community mental health services for people with SMI) 3) Evaluate intervention elements that will enhance sustainable adoption and implementation of community-based mental health care for people with SMI, by carrying out implementation research.

ELIGIBILITY:
Inclusion Criteria:

Adults (ages 18-65), current service users, with severe and enduring mental ill-health, which, for clinical purposes, typically relates to diagnostic categories of bipolar disorder, severe depression, or schizophrenia. We use the following definition for SMI:

* Presence of a psychiatric disorder that requires care and treatment (so, they are NOT in symptom remission)
* Has severe limitations in social and community functioning (i.e. they are not in functional remission)
* These problems are not transient (e.g. temporary, one-off) in nature (They are systematic and long-term)
* Coordinated care provided by care networks or teams is needed to implement the treatment plan

Exclusion Criteria:

Exclusion criteria at the patient level includes patients who do not consent to their data being collected who are part of the intervention or control conditions, those who are under the age of 18 at the start of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in daily functioning | baseline, 12 months, 18 months
  World Health Organisation Disability Assessment Schedule 2 (WHODAS2) measures health and disability-level of functioning in 6 domains:Cognition, Mobility, Self-care,Getting along, Life activities, Participation in community activities.The instrument is self-reporting; can be administered by a health worker if needed. Answers are distributed into 5 categories:"none","mild","moderate","severe"and"extreme or cannot do". It ends with 3 items where answers are presented as number of days (when difficulties were present). Score on any dimension ranges 0 to 7, results are depicted in a diagram which reflects relation between dimensions(the higher the score, the lower level of difficulties/better functioning) and changes over time

SECONDARY OUTCOMES:
Change in health-related quality of life | baseline, 12 months, 18 months
  Euro Quality of Life Index (Euro QoL 5-D 3-L). The instrument measures five dimensions: Mobility, Self-care, Daily activities, Pain/Discomfort and Anxiety/ Depression. Each dimension can be rated at three levels: from no problems to major problems. The five dimensions can be summed into a descriptive health state with 11111 representing no problems in any of the five health dimensions and 33333 indicating major problems in any of the five health dimensions. Second part of the instrument is the Visual Analogue Scale to assess health status at baseline, where 0 signifies worst imaginable health state, and 100 signifies best imaginable health state.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Rojnić Kuzman, A/Prof., Study Chair — Department of Psychiatry
Locations (1):
- KBC Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared with the coordinating institute and Heidelberg University Hospital (two institutions that will be in charge of analyzing data from all participating project sites).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: During the project and for a period of five years after the end of the project; each beneficiary will disseminate its results by disclosing them to the public by appropriate means as soon as possible, including scientific publications in any medium.
Access Criteria: In order to protect participant privacy, data will only be released if the request abides by national and European patient data laws and guidelines, by guidelines for use of mental health data, and by the guidelines set by each research site's ethical review board. Those requesting access to the data will be asked to verify their identity, provide information on how the data will be used, and provide information about their institutions. All requests and releases of data will be logged by the Data Protection Officer. All identifiable data will be kept confidential and will not be released. Data access will be limited to a need only basis. All research partners involved in RECOVER-E will have access to open data sets. As well, datasets will be made available to the European Commission or Global Alliance for Chronic Diseases on request. All de-identified data sets will be stored at the coordinating institute on password-protected, non-networked servers with limited access.

REFERENCES:
- [Derived] Shields-Zeeman L, Smit F, Wijnen B, Roth C, Wensing M, Petrea I; RECOVER-E consortium; Bolinski F, Bajraktarov S, Dedovic J, Keet R, Rojnic Kuzman M, Nakov V, Nica R, Novotni A, Tomcuk A, Djurisic T, Morales G, Rotaru Anghelescu T; RECOVER-E study. Community versus institutionalised care for people with severe mental illness in five countries in Southeast Europe: pooled analysis of five randomised trials. BMJ Glob Health. 2025 Oct 23;10(10):e018594. doi: 10.1136/bmjgh-2024-018594. PMID 41130742
- [Derived] Roth C, Wensing M, Kuzman MR, Bjedov S, Medved S, Istvanovic A, Grbic DS, Simetin IP, Tomcuk A, Dedovic J, Djurisic T, Nica RI, Rotaru T, Novotni A, Bajraktarov S, Milutinovic M, Nakov V, Zarkov Z, Dinolova R, Walters BH, Shields-Zeeman L, Petrea I. Experiences of healthcare staff providing community-based mental healthcare as a multidisciplinary community mental health team in Central and Eastern Europe findings from the RECOVER-E project: an observational intervention study. BMC Psychiatry. 2021 Oct 24;21(1):525. doi: 10.1186/s12888-021-03542-2. PMID 34689733
- [Derived] Wijnen BFM, Smit F, Uhernik AI, Istvanovic A, Dedovic J, Dinolova R, Nica R, Velickovski R, Wensing M, Petrea I, Shields-Zeeman L. Sustainability of Community-Based Specialized Mental Health Services in Five European Countries: Protocol for Five Randomized Controlled Trial-Based Health-Economic Evaluations Embedded in the RECOVER-E Program. JMIR Res Protoc. 2020 Jun 1;9(6):e17454. doi: 10.2196/17454. PMID 32476658
- [Derived] Shields-Zeeman L, Petrea I, Smit F, Walters BH, Dedovic J, Kuzman MR, Nakov V, Nica R, Novotni A, Roth C, Tomcuk A, Wijnen BFM, Wensing M. Towards community-based and recovery-oriented care for severe mental disorders in Southern and Eastern Europe: aims and design of a multi-country implementation and evaluation study (RECOVER-E). Int J Ment Health Syst. 2020 Apr 22;14:30. doi: 10.1186/s13033-020-00361-y. eCollection 2020. PMID 32336984